CLINICAL TRIAL: NCT04129710
Title: An Open-label, Multicenter,Randomized Phase 2 Trial to Compare the Efficacy and Safety of Ibrutinib Versus Lenalidomide in Combination With MRE(Methotrexate,Rituximab,Etoposide)-Chemotherapy for Adult Patients With Recurrent/Refractory Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: A Trial to Compare Ibrutinib Versus Lenalidomide in Combination With MRE-chemotherapy for Adult Patients With Recurrent/Refractory Primary Central Nervous System Lymphoma (PCNSL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ruijin Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Fujian Medical University Union Hospital (Other); RenJi Hospital (Other); Shanghai Tong Ren Hospital (Other); Shandong Provincial Hospital (Other Government); Cancer Hospital of Guangxi Medical University (Other); Sir Run Run Shaw Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Yinzhou Hospital Affiliated to Medical School of Ningbo University (Other); Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I2019001413
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-01

CONDITIONS: Recurrent/RefractoryPrimary Central Nervous System Lymphoma (PCNSL)
MeSH Terms: conditions — Recurrence | interventions — ibrutinib; Lenalidomide; Methotrexate; Rituximab; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I-MRE (Experimental): Ibrutinib 560 mg/day daily (starting dose) between days 4 and 28 of each cycle for six cycles. Then Ibrutinib is continued until disease progression, intolerable toxicity, death or up to two years.
  Methotrexate (standard hydration/leucovorin support) 3.5 g/m2 (0.5 g/m2 in 15 min+ 3 g/m2 in 3-hr infusion) d2.
  Rituximab 375 mg/m2 conventional infusion d1.Etoposide 250 mg/m2 over 3 hours on day3.
  Every 4 weeks for 1 cycle, 6 cycles will be prescribed as protocol.
  Interventions: Drug: Ibrutinib; Drug: Methotrexate; Drug: Rituximab; Drug: Etoposide; Drug: PEGylated recombinant human granulocyte colony
- L-MRE (Experimental): Oral lenalidomide 25mg/day (starting dose) between days 4 and 24 of each cycle for six cycles.Then lenalidomide is continued until disease progression, intolerable toxicity, death or up to two years.
  Methotrexate (standard hydration/leucovorin support) 3.5 g/m2 (0.5 g/m2 in 15 min+ 3 g/m2 in 3-hr infusion) d2.
  Rituximab 375 mg/m2 conventional infusion d1.
  Etoposide 250 mg/m2 over 3 hours on day3.
  Every 4 weeks for 1 cycle, 6 cycles will be prescribed as protocol.
  Interventions: Drug: Lenalidomide; Drug: Methotrexate; Drug: Rituximab; Drug: Etoposide; Drug: PEGylated recombinant human granulocyte colony
- MRE (Active Comparator): Methotrexate (standard hydration/leucovorin support) 3.5 g/m2 (0.5 g/m2 in 15 min+ 3 g/m2 in 3-hr infusion) d2.
  Rituximab 375 mg/m2 conventional infusion d1.
  Etoposide 250 mg/m2 over 3 hours on day3.
  Every 4 weeks for 1 cycle, 6 cycles will be prescribed as protocol.
  Patients who will not achieve SD or better after the 4th course, as well as those who will experience Progressive Disease (PD) at any time will be randomly allocated to the Experimental groups.
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: Etoposide; Drug: PEGylated recombinant human granulocyte colony

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 560 mg/day daily (starting dose) between days 4 and 28 of each cycle for six cycles. Then Ibrutinib is continued until disease progression, intolerable toxicity, death or up to two years.
  Arms: I-MRE
Drug: Lenalidomide — Oral lenalidomide 25mg/day between days 4 and 24 of each cycle for six cycles. Then lenalidomide is continued until disease progression, intolerable toxicity, death or up to two years.
  Arms: L-MRE
Drug: Methotrexate — Methotrexate 3.5 g/m2 (0.5 g/m2 in 15 min + 3 g/m2 in 3-hr infusion) on day 1
Drug: Rituximab — Rituximab 375 mg/m2 conventional infusion on day 1
Drug: Etoposide — Etoposide 250 mg/m2 over 3 hours on day3
Drug: PEGylated recombinant human granulocyte colony — PEGylated recombinant human granulocyte colony 100 ug/kg subcutaneous injection on day 5.

SUMMARY:
This is a open-label，multicenter, randomised, three-arm, phase II efficacy and safety study of ibrutinib in combination with MRE(methotrexate,rituximab,etoposide)-chemotherapy versus lenalidomide in combination with MRE-chemotherapy given to adult patients who have recurrent/refractory primary central nervous system lymphoma (PCNSL)

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to understand and be willing to sign a written informed consent document.
2. Men and woman who are 18-75 years old on the day of consenting to the study.
3. Histologically documented PCNSL and histologically documented systemic diffuse large B-cell lymphoma (DLBCL).
4. Patients must have relapsed/refractory PCNSL or relapsed/refractory SCNSL
5. All patients need to have received at least one prior CNS directed therapy. There is no restriction on the number of recurrences.
6. Patients with parenchymal lesions must have unequivocal evidence of disease progression on imaging (MRI of the brain or head CT) 21 days prior to study registration.
7. Participants must have an ECOG performance status of 0-3.
8. Participants must have adequate bone marrow and organ function shown by:

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
   2. Platelets ≥ 75 x 10^9/L and no platelet transfusion within the past 21 days prior to study registration
   3. Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 21 days prior to study registration
   4. International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
   6. Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome.
   7. Serum creatinine ≤ 2 times the upper limit of normal
9. Woman of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose.
10. Patients must be able to tolerate MRI/CT scans.
11. Participants must have recovered to grade 1 toxicity from prior therapy.
12. Participants should be able to submit up to 20 unstained formalin-fixed, paraffinembedded (FFPE) slides from the initial tissue diagnosis prior to study registration for confirmation of diagnosis and correlative studies
13. NOTE: Prior autologous stem cell transplant as well as prior radiation to the CNS does NOT prevent patients from enrollment into the trial.

Exclusion Criteria:

1. Patients with SCNSL actively receiving treatment for extra-CNS disease are excluded.
2. Patient has received chemotherapy, monoclonal antibodies or targeted anticancer therapy ≤ 4 weeks or 5 half-lives, whichever is shorter, or 6 weeks for nitrosourea or mitomycin-C prior to starting the study drug, or the patient has not recovered from the side effects of such therapy.
3. Patient has received external beam radiation therapy to the CNS within 21 days of the first dose of the study drug.
4. Patient requires more than 8 mg of dexamethasone daily or the equivalent
5. Patient has an active concurrent malignancy requiring active therapy
6. The patient has been treated with radio- or toxin-immunoconjugates within 70 days of the first Patient is allergic to components of the study drug.
7. Patient is using warfarin or any other Coumadin-derivative anticoagulant or vitamin K antagonists. Patients must be off warfarin-derivative anticoagulants for at least seven days prior to starting the study drug. Low molecular weight heparin is allowed. Patients with congenital bleeding diathesis are excluded.
8. Patient is taking a drug known to be a moderate and strong inhibitor or inducers of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers for at least two weeks prior to starting the study drug.
9. Patient is using systemic immunosuppressant therapy, including cyclosporine A, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day or prednisone or the equivalent. Participants must be off immunosuppressant therapy for at least 28 days prior to the first dose of the study drug.
10. Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening,
11. Patient has a known bleeding diathesis (e.g. von Willebrand"s disease) or hemophilia.
12. Patient is known to have human immunodeficiency virus (HIV) infection.
13. Patient is known to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests.
14. Patient is known to have an uncontrolled active systemic infection.
15. Patient underwent major systemic surgery ≤ 4 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery, or who plan to have surgery within 2 weeks of the first dose of the study drug.
16. Patient is unable to swallow capsules or has a disease or condition significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction.
17. Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject"s safety or put the study outcomes at undue risk.
18. Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive serum hCG laboratory test of > 5 mIU/mL (See section on Pregnancy and Reproduction)
19. Patient has undergone prior allogenic stem cell transplant (autologous stem cell transplant is NOT an exclusion)
20. The patient is unwell or unable to participate in all required study evaluations and procedures
21. Known hypersensitivity to ibrutinib, thalidomide or lenalidomide

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | assessed up to 2 yrs
  From date of randomization until recurrence/disease progression, unacceptable toxicity, death or discontinuation for any other reason, whichever comes first assessed up to 2 yrs

SECONDARY OUTCOMES:
Objective response rate (ORR) | assessed up to 2 yrs
  To determine efficacy
Overall survival (OS) | assessed up to 2 yrs
  To determine efficacy
Number of patients with adverse events | assessed up to 2 yrs
  Number of participants with treatment- and non-treatment related adverse events as assessed by CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China/Zhejiang Province, China

IPD SHARING:
Plan to Share IPD: Yes
This is a open-label，multicenter, randomised, three-arm, phase II efficacy and safety study of ibrutinib in combination with MRE(methotrexate,rituximab,etoposide)-chemotherapy versus lenalidomide in combination with MRE-chemotherapy given to adult patients who have recurrent/refractory primary central nervous system lymphoma (PCNSL)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code